CLINICAL TRIAL: NCT03398473
Title: A Phase 1, Open-label, Randomized, Single Dose, Crossover Study Evaluating The Pharmacokinetics Of Epoetin Following Administration Of Epoetin Hospira Multiple Dose Vial (Mdv) Product Compared To Epoetin Hospira Single Dose Vial (Sdv) Product As Subcutaneous Injection To Normal Healthy Subjects
Brief Title: A Study Comparing The Effects Of Epoetin Hospira Single-Dose Vial (SDV) And Multi-Dose Vial (MDV) When Administered Subcutaneously To Normal Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C3461009
Record Dates: First submitted 2018-01-08; First posted 2018-01-12 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: Epoetin Hospira; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Epoetin Hospira SDV (Experimental): Epoetin Hospira Single Dose Vial (SDV)
  Interventions: Drug: Epoetin Hospira SDV
- Epoetin Hospira MDV (Experimental): Epoetin Hospira Multi-Dose Vial (MDV)
  Interventions: Drug: Epoetin Hospira MDV

INTERVENTIONS:
Drug: Epoetin Hospira SDV — Epoetin Hospira Single Dose Vial
  Arms: Epoetin Hospira SDV
Drug: Epoetin Hospira MDV — Epoetin Hospira Multi-Dose Vial
  Arms: Epoetin Hospira MDV

SUMMARY:
This study will assess the PK similarity of epoetin administered as Hospira MDV versus Hospira SDV by conducting a single-dose comparative evaluation in normal healthy subjects enrolled at a single center.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects who, at time of Screening, are between ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure and pulse rate measurement, 12-lead electrocardiogram, or clinical laboratory tests.

   Female subjects of nonchildbearing potential must meet at least 1 of the following criteria:
   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; a serum follicle-stimulating hormone (FSH) level confirming the postmenopausal state.
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure.
2. Body Mass Index of 17.5 to 30.5 kg/m2; and a total body weight > 50 kg (110 lbs).
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
4. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence of history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing), cancer, (except for basal cell carcinoma of skin), erythrocytosis, or seizures.
2. Any condition possibly affecting drug absorption (e.g. gastrectomy).
3. History of bleeding ulcer, bleeding abnormalities or coagulation abnormalities.
4. A positive urine drug screen.
5. Use of tobacco or nicotine-containing products within 3 months of Screening or a positive urine cotinine test (ie, active smokers and those who currently use nicotine-containing products are excluded from participation in this study).
6. Significant drug sensitivity or a significant allergic reaction to any drug, as well as known hypersensitivity or idiosyncratic reaction to epoetin (or its excipients, including benzyl alcohol and any other related drugs).
7. Any previous use of epoetin.
8. History of regular alcohol consumption exceeding 7 drinks/week for female subjects or 14 drinks/week for male subjects (1 drink = 5 oz. [150 mL] of wine or as oz. [360 mL] of beer or 1.5 oz. [45 mL] of hard liquor) within 6 months before Screening.
9. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceeding the fits dose of investigational product (whichever is longer).
10. Screening supine BP >= 140 mmHg (systolic) or >=90 mmHg (Diastolic), following at least 5 minutes of supine rest. If BP >= 140 mmHg (systolic) or >= 90 mmHg (Diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.
11. Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval> 450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
12. Subject's with ANY of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * Aspartate aminotransferase (AST) OR alanine aminotransferase (ALT) leve l>= 1.5 X upper limit of normal (ULN);
    * Total bilirubin level 1.5 X ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <= ULN.
13. Pregnant female subjects; breastfeeding female subjects; fertile male subjects and female subjects of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outline in the protocol for the duration of the study and for at least 30 days after the last dose of investigational product.
14. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product. As exceptions, acetaminophen/paracetamol may be used at doses of <= 1 g/day and hormonal contraceptives will be allowed. Limited use of nonprescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
15. A subject who has been administered a drug by depot injection within 30 days prior to the initial study drug administration or 6 half-lives of that drug, whichever is longer and at the discretion of the investigator, or who has received a recent (6 weeks prior to admission to the CRU) live or attenuated vaccination, or exposure to communicable viral diseases such as chicken pox, varicella, and measles.
16. Blood donation (excluding plasma donations) or approximately 1 pint (500 mL) or more within 60 days prior to dosing.
17. History of HIV, hepatitis B, or hepatitis C, positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
18. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of the protocol.
19. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
20. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgement of the investigator, would make the subject inappropriate for entry into this study.
21. May not be able to comply with the requirements of this clinical trial or be able to communicate effectively with study personnel, or is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration (C max) of PF-06946151 SDV | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96, and 120 hours after dose administration]
Maximum serum concentration (C max) of PF-06946151 MDV | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96, and 120 hours after dose administration]
Area under the serum PF-06946151 SDV concentration-time profile (AUC last) from time 0 to the last quantifiable concentration (C last) | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96, and 120 hours after dose administration]
Area under the serum PF-06946151 MDV concentration-time profile (AUC last) from time 0 to the last quantifiable concentration (C last) | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96, and 120 hours after dose administration]
Area under the PF-06946151 SDV concentration-time profile (AUC inf) from time zero extrapolated to infinity | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96, and 120 hours after dose administration]
Area under the PF-06946151 MDV concentration-time profile (AUC inf) from time zero extrapolated to infinity | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96, and 120 hours after dose administration]

SECONDARY OUTCOMES:
Time to reach maximum concentration (T max) of PF-06946151 SDV | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96 and 120 hours after dose administration]
Time to reach maximum concentration (T max) of PF-06946151 MDV | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96 and 120 hours after dose administration]
Elimination half life (T 1/2) of PF-06946151 SDV | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96 and 120 hours after dose administration]
Elimination half life (T 1/2) of PF-06946151 MDV | [Time Frame: 0, 0.5, 3, 6, 9, 12, 15, 24, 30, 36, 48, 72, 96 and 120 hours after dose administration]
Number of subjects with adverse events (AEs) by severity and relationship to treatment | Day 1 through approximately Day 30 after Period 2
Number of subjects with abnormal physical exam findings | Day 1 through approximately Day 30 after Period 2
Percentage of subjects with the development of Anti-Drug Antibodies | Day 1 through approximately Day 30 after Period 2
Number of subjects with change from baseline in laboratory results | Day 1 through approximately Day 30 after Period 2
Number of subjects with clinically relevant changes in vital signs since baseline | Day 1 through approximately Day 30 after Period 2
Percentage of subjects with the development of Neutralizing Antibodies | Day 1 through approximately Day 30 after Period 2

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C3461009&StudyName=A+Phase+1%2C+Open-label%2C+Randomized%2C+Single+Dose%2C+Crossover+Study+Evaluating+The+Pharmacokinetics+Of+Epoetin+Following+Administration+Of+Epoetin+Hospira+Multiple+Dose+Vial+%28mdv%29+Product+Compared+To+Epoetin+Hospira+Single+Dose+Vial+%28sdv%29+Product+As+Subcutaneous+Injection+To+Normal+Healthy+Subjects